CLINICAL TRIAL: NCT06488248
Title: Endoscopic Third Ventriculostomy Compared to Ventriculoperitoneal Shunt as Treatment for Idiopathic Normal Pressure Hydrocephalus (ENDOVEST): A Randomized Trial
Brief Title: Endoscopic Third Ventriculostomy vs. Ventriculoperitoneal Shunt in Idiopathic Normal Pressure Hydrocephalus (ENDOVEST)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-00845; ko23Soleman
Record Dates: First submitted 2024-06-18; First posted 2024-07-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus (INPH)
Keywords: Surgical treatment; Neurosurgery; Endoscopic third ventriculostomy (ETV); Ventriculoperitoneal shunt (VPS)
MeSH Terms: interventions — Ventriculostomy; Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic third ventriculostomy (ETV) group (Experimental): The investigational group undergoes endoscopic third ventriculostomy (ETV) for the treatment of idiopathic normal pressure hydrocephalus (iNPH).
  Interventions: Procedure: Endoscopic third ventriculostomy (ETV)
- Ventriculoperitoneal shunt (VPS) group (Other): The control group undergoes ventriculoperitoneal shunt (VPS) implantation for the treatment of iNPH.
  Interventions: Procedure: Ventriculoperitoneal shunt (VPS)

INTERVENTIONS:
Procedure: Endoscopic third ventriculostomy (ETV) — The procedure is performed using an endoscope (LOTTA® system, Karl Storz Endoscopes, Germany; Minop®, BBraun, Tuttlingen, Germany or equivalent). The intervention is carried out under general anesthesia, with the procedure typically lasting around 60 minutes.
  Arms: Endoscopic third ventriculostomy (ETV) group
Procedure: Ventriculoperitoneal shunt (VPS) — The procedure entails the insertion of a catheter into both the ventricular system and the peritoneal cavity, connected to a programmable valve that regulates cerebrospinal fluid flow. The choice of programmable valve (Codman Hakim or Codman Certas Programmable Valves, Integra, Plainsboro, USA; Strata valve, Medtronic, Minneapolis, USA; Sophysa, Orsay, France; Miethke proGAV, Aesculap, Tuttlingen, Germany) is at the surgeon's discretion. The preoperative valve setting is preset to a pressure level between 85 - 135 mmH2O. The VPS procedure is conducted under general anesthesia and typically lasts approximately 90-120 minutes.
  Arms: Ventriculoperitoneal shunt (VPS) group

SUMMARY:
The aim of this single-center, two-arm, open-labeled, randomized controlled clinical study is to compare two surgical interventions, endoscopic third ventriculostomy and ventriculoperitoneal shunt, in treating idiopathic normal pressure hydrocephalus in terms of clinical improvement.

DETAILED DESCRIPTION:
Idiopathic normal pressure hydrocephalus (iNPH) primarily affects elderly individuals, with prevalence rates of approximately 1.4% among those over 65 years and 5.9% among those over 80 years old. It is characterized by fluid buildup in the brain with normal cerebrospinal fluid pressure and is unique among neurodegenerative disorders in its potential for successful treatment. Common symptoms include difficulty walking, urinary incontinence, and cognitive decline, which significantly impact quality of life.

The standard treatment involves inserting a ventriculoperitoneal shunt (VPS) to drain cerebrospinal fluid, achieving a 75% success rate in improving symptoms. However, VPS has a drawback: a high rate of revision surgery (approximately 18% during follow-up). An alternative treatment is endoscopic third ventriculostomy (ETV), which avoids placing foreign materials and thus eliminates risks associated with shunt malfunction and infections. ETV is an established neuroendoscopic procedure mainly used to treat non-communicating hydrocephalus, typically due to aqueduct stenosis.

This study aims to compare ETV and VPS for the treatment of iNPH to investigate whether ETV leads to fewer complications while achieving a comparable rate of postoperative symptom improvement.

ELIGIBILITY:
Inclusion Criteria:

* >40 years of age
* Symptom duration ≥3 months, <24 months
* No antecedent head trauma, ICH, meningitis, or other cause of secondary hydrocephalus
* MUST show gait/balance disturbance, PLUS cognition impairment AND/OR urinary dysfunction.
* Ventricular enlargement (Evans Index > 0.3) not attributable to cerebral atrophy or congenital enlargement
* No macroscopic obstruction to cerebrospinal fluid (CSF) flow Spinal Tap-Test
* Opening pressure (on lateral decubitus): <24cmH2O
* Clinical improvement in at least one of the main symptoms after 40-50ml withdrawal of CSF

Exclusion Criteria:

* ≤40 years of age
* No informed consent
* Other neurologic, psychiatric or general medical condition which is sufficient to explain the presenting symptoms.
* Previous cranial neurosurgical interventions
* Other associated dementia syndromes
* Incapacity to walk
* Pregnancy and breastfeeding women

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
idiopathic normal pressure hydrocephalus (iNPH) score | Before surgery (baseline), up to 5 days, 2, 6, and 12 months after surgery
  The idiopathic normal pressure hydrocephalus (iNPH) score is used to measure the clinical improvement and complication rate. The iNPH score evaluates the three cardinal symptoms of iNPH-gait disturbance, dementia, and urinary incontinence-with each category assigned a score between 0 and 4 based on severity, resulting in a total score ranging from 0 (indicating normal) to 12 (reflecting the maximum severity of symptoms The score will be assessed during the outpatient consultation before surgery, at admission directly preceding surgery, and postoperatively at discharge, as well as during follow-up at 6-8 weeks, 6 months, and 12 months after the operation.

SECONDARY OUTCOMES:
Level of consciousness (Glasgow Coma Scale) | Before surgery (baseline), up to 5 days, 2, 6, and 12 months after surgery
  The Glasgow Coma Scale (GCS) is used to assess the level of consciousness by evaluating eye, verbal, and motor responses. The GCS score ranges from 3 to 15, with higher scores indicating better neurological function and a less severe brain injury. A score of 3 represents deep unconsciousness, while a score of 15 indicates full alertness and orientation.
Degree of disability and dependency (modified Rankin Scale) | Up to 5 days, 2, 6, and 12 months after surgery
  The modified Rankin Scale (mRS) is used to assess the degree of disability and dependency in everyday life. Th mRS is a standard tool to assess the neurological outcome in trials with acute severe brain disease. The mRS ranges from 0 (no disability) to 6 (death). Lower values indicate less disability.
Cognitive function (Montreal Cognitive Assessment) | Before surgery (baseline), up to 5 days, 2, 6, and 12 months after surgery
  The Montreal Cognitive Assessment (MoCA) is used to evaluate cognitive function and detect mild cognitive impairment. It scores between 0 and 30, with higher scores indicating better cognitive performance. A score of 26 or above is generally considered normal.
GaitRite walkway | At 2 and 12 months after surgery
  To assess the gait and balance, a 10-metre GaitRite walkway, specifically designed to measure and analyze gait patterns, is performed. The body's movement are recorded using the the Ambulatory Parkinson's Disease Monitoring (APDM) Mobility Lab System.
Timed-Up-and-Go Test | At 2 and 12 months after surgery
  To assess the gait and balance, the Timed-Up-and-Go Test is performed. This is a simple and quick assessment to measure the time taken for an individual to stand up from a chair, walk three meters, turn around, walk back to the chair, and sit down again, with shorter times indicating better mobility.
Modified Clinical Test of Sensory Interaction on Balance | At 2 and 12 months after surgery
  To assess the gait and balance, the modified Clinical Test of Sensory Interaction on Balance (mCTSIB, 30 seconds) is performed. The mCTSIB measures a person's ability to maintain stability in different sensory conditions for 30 seconds each.
Modified Balance Error Scoring System | Before surgery (baseline), at 2 and 12 months after surgery
  To assess the gait and balance, the modified Balance Error Scoring System (mBESS) is performed. The mBESS involves performing three standing balance tasks (double-leg stance, single-leg stance, and tandem stance) on both firm and foam surfaces, with errors recorded to gauge balance performance.
5-times-sit-to-stand test | At 2 and 12 months after surgery
  To assess the gait and balance, the 5-times-sit-to-stand test is performed. It involves timing how long it takes a person to rise from a seated position to a standing position five times as quickly as possible.
Hand grip strength test | At 2 and 12 months after surgery
  To assess the gait and balance, the hand grip strength test is performed. It assesses the maximum isometric strength of the hand and forearm muscles and involves using a dynamometer to measure the force exerted when a person squeezes the device with their hand.
Montreal Cognitive Assessment | At 2 and 12 months after surgery
  As a neuropsychological assessment the Montreal Cognitive Assessment is performed to evaluate cognitive function and detect mild cognitive impairment. It assesses various cognitive domains, including memory, attention, language, and executive functions, with a maximum score of 30 points; higher scores indicate better cognitive function.
Test of Attentional Performance | At 2 and 12 months after surgery
  As a neuropsychological assessment the TAP Test (Test of Attentional Performance) is a computer-based assessment used to evaluate different aspects of attention, such as alertness, divided attention, and sustained attention. It measures reaction times and accuracy across various tasks designed to assess cognitive functions related to attentional control and processing speed.
Trail Making Test | At 2 and 12 months after surgery
  As a neuropsychological assessment the Trail Making Test is performed to evaluate cognitive flexibility, visual attention, and task-switching abilities. It consists of two parts: Part A involves connecting numbered circles sequentially, while Part B requires alternating between numbers and letters in ascending order. The test measures executive functioning and processing speed, with longer completion times indicating potential cognitive impairment.
Stroop-Test | At 2 and 12 months after surgery
  As a neuropsychological assessment the Stroop-Test is performed to measure selective attention, cognitive flexibility, and processing speed. It typically involves presenting color names (e.g., "red," "blue") printed in incongruent colored ink (e.g., the word "red" printed in blue ink), and participants are required to name the ink color while ignoring the word. The test assesses the ability to inhibit automatic responses and is sensitive to cognitive impairments, with longer response times or increased errors indicating potential difficulties in executive functioning.
CERAD Word List | At 2 and 12 months after surgery
  The Consortium to Establish a Registry for Alzheimer's Disease (CERAD) Word List is used as a neuropsychological assessment to evaluate verbal memory. It consists of a list of 10 common words that the participant is asked to recall immediately after hearing them. This test assesses the ability to remember and retrieve information shortly after it was presented, providing insights into memory function and potential cognitive impairments.
CERAD Constructive Praxis | At 2 and 12 months after surgery
  The CERAD Constructive Praxis is used as a neuropsychological assessment to assess visuospatial and constructional abilities by asking participants to copy a series of geometric figures. This test helps evaluate visual perception, spatial orientation, and motor skills, providing insights into cognitive functioning.
Boston Naming Test | At 2 and 12 months after surgery
  As a neuropsychological assessment the Boston Naming Test is performed. It assesses the ability to name objects or pictures presented by the examiner, evaluating language and semantic memory functions.
Rey-Osterrieth Complex Figure Test | At 2 and 12 months after surgery
  As a neuropsychological assessment the Rey-Osterrieth Complex Figure Test is performed. It assesses visuospatial and constructional abilities as well as visual memory. It involves copying a complex figure and then recalling and reproducing it from memory.
Intensity of depression (Beck Depression Inventory) | Before surgery (baseline), at 2 and 12 months after surgery
  The Beck Depression Inventory (BDI) is used to assess the intensity of depression. The BDI is a self-report questionnaire designed to assess the severity of depressive symptoms. It consists of 21 multiple-choice questions, each related to a specific symptom of depression such as sadness, pessimism, guilt, and fatigue. Scores on the BDI can range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Flow-void presence | Up to 5 days, 2, 6, and 12 months after surgery
  In a radiological assessment the flow-void presence is determined.
Ventricular volumetry | Up to 5 days, 2, 6, and 12 months after surgery
  In a radiological assessment the ventricular volumetry is measured.
Periventricular perfusion measurements | Up to 5 days, 2, 6, and 12 months after surgery
  In a radiological assessment periventricular perfusion measurements are carried out.
iNPH Radiological Scale | Up to 5 days, 2, 6, and 12 months after surgery
  In a radiological assessment the idiopathic normal pressure hydrocephalus (iNPH) radiological scale is assessed. Scores typically range from 0 to 12, with higher scores indicating greater severity of radiological findings suggestive of iNPH, such as enlarged ventricles, narrow sulci, and periventricular white matter changes.
iNPH severity | Before surgery (baseline), up to 5 days, 2, 6, and 12 months after surgery
  iNPH severity is measured using the Hellström score, which ranges from 0 to 12, with higher scores indicating more severe symptoms across domains of gait, balance, and cognitive impairment.
Health-related quality of life | At 2, 6, and 12 months after surgery
  The quality of life is assessed using the 15D health-related quality of life (HRQoL) patient-reported questionnaire. It cover aspects like physical functioning, emotional well-being, social functioning, and pain. Scores can range from 0 to 100, with higher scores reflecting better perceived health and functioning across various domains, while lower scores suggest greater impairment and reduced quality of life.
Evaluation of complications | Up to 5 days, 2, 6, and 12 months after surgery
  During hospitalization, 6-8 weeks, as well as 6- and 12-month follow-up, the incidence of complications is assessed. Complications are defined as infections, bleeding, shunt dysfunction (e.g., due to misplacement, obstruction of the proximal ventricular catheter, dysfunction of the valve, dysfunction of the peritoneal catheter), ETV occlusions (requiring re-ETV or VPS insertion), and neuronal tissue injury (e.g., fornix injury).
Evaluation of revision surgery | Up to 5 days, 2, 6, and 12 months after surgery
  during hospitalization, 6-8 weeks, as well as 6- and 12-month follow-up, the incidence and reason of revision surgery is assessed.
Mortality | Up to 5 days, 2, 6, and 12 months after surgery
  The mortality is assessed during hospitalization and the 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Florian Marc Ebel, Dr. med., Principal Investigator — Department of Neurosurgery, University Hospital of Basel
Locations (1):
- Department of Neurosurgery, University Hospital of Basel, Basel, Switzerland